CLINICAL TRIAL: NCT06698640
Title: Optimization of HEDIS Gap Closure Strategies for Well-Child Visits: A Three-Arm Randomized Controlled Trial
Brief Title: A Trial of Text-Message-Based Engagement for Well-Child Visits
Acronym: HEDIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Waymark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HEDIS-OPT-2024-001
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Well Child Visit; Gaps in Care
Keywords: gaps in care; preventive care; text messaging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will receive traditional passive outreach, which includes standard reminders and communications that do not utilize automated technologies.
- Automated SMS (Active Comparator): Participants will receive automated SMS messages reminding them of their Well-Child Visits. These messages will be standardized and sent at intervals designed to prompt appointment attendance.
  Interventions: Behavioral: Automated SMS
- Automated SMS + Scheduling Assistance (Active Comparator): Participants will receive the same automated SMS messages as in Arm 2, but with the added component of proactive appointment scheduling assistance. This may include options for scheduling directly through the SMS platform or follow-up messages encouraging appointment setting.
  Interventions: Behavioral: Automated SMS + Scheduling Assistance

INTERVENTIONS:
Behavioral: Automated SMS — Participants will receive automated SMS messages reminding them of their Well-Child Visits. These messages will be standardized and sent at intervals designed to prompt appointment attendance.
  Arms: Automated SMS
Behavioral: Automated SMS + Scheduling Assistance — Participants will receive the same automated SMS messages as in Arm 2, but with the added component of proactive appointment scheduling assistance. This may include options for scheduling directly through the SMS platform or follow-up messages encouraging appointment setting.
  Arms: Automated SMS + Scheduling Assistance

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of different outreach strategies in closing HEDIS gaps for Well-Child Visits (WCV) in children aged 0-21 years. The main questions it aims to answer are:

Does automated SMS outreach improve the rate of completed Well-Child Visits compared to traditional passive outreach? Does the combination of automated SMS and appointment scheduling assistance lead to higher completion rates than automated SMS alone?

Researchers will compare three groups to see if the different outreach strategies have varying effects on WCV completion rates:

Control Group: Participants will receive traditional passive outreach (current standard practice).

Automated SMS Group: Participants will receive standardized SMS messages to remind them of their Well-Child Visits.

Automated SMS + Scheduling Assistance Group: Participants will receive SMS messages along with proactive assistance in scheduling their appointments.

Participants will:

Be randomized into one of the three study groups. Receive outreach according to their group assignment. Have their appointment scheduling and attendance tracked. Contribute data that will help evaluate the effectiveness of each outreach strategy in closing HEDIS gaps for Well-Child Visits.

This study aims to optimize outreach methods to improve healthcare delivery and preventive care adherence for pediatric populations.

DETAILED DESCRIPTION:
Study Overview:

This clinical trial aims to evaluate the effectiveness of different outreach strategies in closing Healthcare Effectiveness Data and Information Set (HEDIS) gaps for Well-Child Visits (WCV) among children aged 0-21 years. HEDIS measures are critical indicators of healthcare quality and preventive care adherence, and improving outreach methods is essential for enhancing healthcare delivery systems.

Purpose of the Study:

The primary purpose of this study is to determine if automated outreach methods, specifically automated Short Message Service (SMS) communications, can effectively increase the rates of completed Well-Child Visits compared to traditional passive outreach methods. The study also aims to evaluate the added benefit of integrating appointment scheduling assistance with automated SMS reminders.

Research Questions:

The main questions this study aims to answer are:

Does automated SMS outreach improve the rate of completed Well-Child Visits compared to traditional passive outreach? Does the combination of automated SMS and appointment scheduling assistance lead to higher completion rates than automated SMS alone?

Study Design:

This is a three-arm randomized controlled trial. Participants will be randomly assigned to one of the following three groups:

Arm 1 (Control): Participants will receive traditional passive outreach, which includes standard reminders and communications that do not utilize automated technologies.

Arm 2 (Automated SMS): Participants will receive automated SMS messages reminding them of their Well-Child Visits. These messages will be standardized and sent at intervals designed to prompt appointment attendance.

Arm 3 (Automated SMS + Scheduling Assistance): Participants will receive the same automated SMS messages as in Arm 2, but with the added component of proactive appointment scheduling assistance. This may include options for scheduling directly through the SMS platform or follow-up messages encouraging appointment setting.

Participant Population:

The study will enroll 180 subjects who have not conducted their recommended Well-Child Visits. Each arm will consist of 60 participants. The study will focus on parents or guardians of children who have an open HEDIS gap for Well-Child Visits at the start of the study.

Inclusion Criteria:

Participants must meet the following criteria:

Have an open HEDIS gap for Well-Child Visits at the start of the study. Be part of the patient list from which Waymark is authorized to conduct outreach.

Have valid contact information, including a phone number capable of receiving SMS.

Exclusion Criteria:

Participants will be excluded if they:

Have opted out of receiving SMS communications. Lack the ability to receive SMS messages. Have requested no contact from their healthcare provider or health plan.

Study Procedures:

Identification of Eligible Patients: Eligible patients with open HEDIS gaps for Well-Child Visits will be identified from existing patient lists.

Randomization: Patients will be randomly assigned to one of the three study arms.

Implementation of Outreach Strategy:

Arm 1 will continue with no changes to current practice. Arm 2 will involve sending standardized SMS messages to remind participants of their Well-Child Visits.

Arm 3 will include sending SMS messages along with proactive scheduling assistance.

Tracking Outcomes: Appointment scheduling and attendance will be monitored, and data on HEDIS gap closure rates will be collected.

Data Collection: Information on staff time and resources used for each intervention will also be collected to evaluate efficiency.

Outcome Measures:

Primary Outcome: The primary outcome will be the rate of HEDIS gaps closed per week/month for each arm.

Secondary Outcome: The secondary outcome will assess the staff time (in minutes) required per gap closure.

Tertiary Outcome: For Arm 3 only, the percentage of automated scheduling attempts requiring human intervention will be documented.

Data Analysis:

Statistical analyses will be conducted to compare outcomes across the three arms using appropriate methods, such as ANOVA and chi-square tests. Subgroup analyses will be performed separately for Well-Child Visits to understand the effectiveness of the interventions within this specific population.

Data Monitoring and Confidentiality:

Data will be stored on secure, HIPAA-compliant servers with encryption. Access will be limited to authorized personnel. De-identified data will be used for analysis wherever possible, and a secure key linking study IDs to patient identifiers will be maintained separately.

Risk/Benefit Assessment:

This study is categorized as minimal risk. Potential risks include:

Privacy breaches (minimal likelihood due to robust data security measures). Patient annoyance with SMS messages (participants can opt-out). Miscommunication of appointment details (verification steps included).

Potential Benefits:

Increased likelihood of receiving timely preventive care. Convenient appointment scheduling for participants in Arm 3. Improved health outcomes associated with closing HEDIS gaps.

Subject Recruitment and Consent:

Subjects will be identified from existing patient lists where Waymark is authorized to conduct outreach. The study requests a waiver of informed consent due to the minimal risk involved and the nature of the interventions, which are variations of standard practices.

Conclusion:

This study aims to provide valuable insights into the effectiveness of automated outreach strategies in improving Well-Child Visit completion rates. By leveraging existing authorized outreach practices and implementing robust data protection measures, we seek to enhance healthcare delivery systems and contribute to better health outcomes for pediatric populations. The requested waivers of consent and authorization are essential for maintaining the scientific integrity of the study and ensuring meaningful results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 0-21 years old who have not had a pediatric well-child visit in the past year
2. Patients for whom the care team is authorized to conduct outreach per the patient's Medicaid health plan
3. Patients with a phone number in health plan eligibility file

Exclusion Criteria:

1. Patients who have opted out of receiving text/SMS communications
2. Patients without the ability to receive text/SMS messages due to lack of valid phone number or active phone
3. Patients who have requested no contact from their healthcare provider or health plan

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2821 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Well child visits attended per month | Monthly for six months of post-intervention observation
  Number of well child visits attended per month

SECONDARY OUTCOMES:
Staff time required per gap closure | Minutes per patient during 6 month observation period
  Minutes spent by staff member per well child visit outreach, engagement, and scheduling tasks
Human escalation rate | Percent of attempts during six months of post-intervention observation
  Percentage of automated scheduling attempts requiring human intervention (Arm 3 only)

CONTACTS AND LOCATIONS:
Locations (1):
- Waymark, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No